CLINICAL TRIAL: NCT02316574
Title: The Role of Neural Systems for Emotion Regulation in Coping With Alcohol Craving
Acronym: FRAME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Nasir Naqvi, research psychiatrist, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: #6859
Record Dates: First submitted 2014-12-10; First posted 2014-12-15 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Alcoholism
Keywords: Alcohol dependence; Cognitive Behavioral Therapy; Functional neuroimaging
MeSH Terms: conditions — Alcoholism | interventions — Cognitive Behavioral Therapy; Secondary Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cognitive Behavioral Coping Skills (Experimental): Cognitive Behavioral Coping Skills Therapy is an individual psychotherapy for alcohol use disorders that has been previously shown to reduce drinking. The focus of this treatment is the teaching of coping skills for managing alcohol craving and negative emotions as a way to reduce drinking behavior.
  Interventions: Behavioral: Cognitive Behavioral Coping Skills Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Coping Skills Therapy — Cognitive Behavioral Coping Skills Therapy (CBCST) is an individual psychotherapy for alcohol dependence that helps individuals to reduce drinking by addressing the ability to regulate, or "cope" with alcohol cravings and other emotions that promote alcohol use.
  Other Names: Cognitive Behavioral Therapy; Relapse Prevention Therapy

SUMMARY:
Cognitive Behavioral Coping Skills Therapy (CBCST) is a commonly utilized, evidence-based psychosocial therapy (talk therapy) for alcohol dependence. By identifying the neural mechanisms through which CBCST changes drinking behavior, it may be possible to improve its efficacy. CBCST promotes abstinence by teaching "coping skills" for managing alcohol-related thoughts and emotions. In this pilot study, the investigators examine the neural systems that play a role in the learning of coping skills through CBCST, specifically focusing on the role of emotion regulation systems.

DETAILED DESCRIPTION:
The study combines 1) a 12-week clinical trial of CBCST in currently drinking alcohol dependent patients (target N=25) who are seeking treatment to reduce their drinking with 2) functional magnetic resonance imaging (fMRI) experiments that probe neural activity related to the utilization of copings skills taught in CBCST. The fMRI studies will be performed both before and after treatment with CBCST, with the goal of determining 1) the pattern of neural activity that is related to coping skills utilization prior to undergoing CBCST, with particular focus on neural systems known to play a role in emotion regulation; 2) how CBCST changes this pattern of neural activity; and 3) how these changes in neural activity predict changes in alcohol use during CBCST.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* Meets DSM-V criteria for current Alcohol Use Disorder
* Currently drinking >5/4 or more drinks/day for men/women in the last 28 day, on average, at the time of initial screening visit.
* Current goal of moderating or abstaining from drinking alcohol
* Seeking treatment for Alcohol Use Disorder
* Agree to not seek additional treatment, apart from Alcoholics Anonymous
* English-speaking and able to provide informed consent and comply with study procedures
* Willing to abstain from alcohol completely for 24 hours on 3 separate occasions

Exclusion Criteria:

* Any current Moderate or Severe substance use disorder, other than alcohol, nicotine or caffeine use disorders.
* Lifetime history of Bipolar Disorder, Schizophrenia or Schizoaffective Disorder
* A diagnosis of any current psychiatric disorder other than Alcohol Use Disorder (e.g. Major Depressive Disorder, Generalized Anxiety Disorder) that in the investigator's judgment might require intervention with either pharmacological or non-pharmacological therapy over the course of the study.
* History of severe alcohol withdrawal (e.g. seizure, delirium tremens, multiple detoxifications or ER visits for alcohol withdrawal)
* Significant risk for suicide or violence
* Legally mandated to receive treatment
* Sufficiently socially unstable as to preclude study participation (e.g. homeless).
* Currently taking any psychotropic medications.
* Significant cognitive impairment
* Neurological or medical conditions that would interfere with MRI scanning (e.g. history of stroke, seizure, brain tumor, brain infection, multiple sclerosis, metal device in body, pregnancy, claustrophobia)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Percent heavy drinking days | 12 weeks
  Assessed during the weekly CBCST treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nasir H. Naqvi, MD, PhD, Principal Investigator — Assistant Professor of Pscyhiatry
Locations (1):
- NYPInstitute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Srivastava AB, Sanchez-Pena J, Levin FR, Mariani JJ, Patel GH, Naqvi NH. Drinking reduction during cognitive behavioral therapy for alcohol use disorder is associated with a reduction in anterior insula-bed nucleus of the stria terminalis resting-state functional connectivity. Alcohol Clin Exp Res. 2021 Aug;45(8):1596-1606. doi: 10.1111/acer.14661. Epub 2021 Aug 2. PMID 34342012